CLINICAL TRIAL: NCT00156299
Title: A Pilot Study of Nuclear Factor-kappa B (NFkB) Inhibition During Induction Chemotherapy for Patients With Acute Myelogenous Leukemia (AML)
Brief Title: Gene Expression During Chemotherapy in Patients With Newly Diagnosed Acute Myeloid Leukemia Treated With Choline Magnesium Trisalicylate
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Replaced by another study
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540303; P30CA072720 (NIH); 020201 (Other: CINJ)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Leukemia
Keywords: adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — choline magnesium trisalicylate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone plus Choline Magnesium Trisalicylate (Experimental): Dexamethasone plus Choline Magnesium Trisalicylate
  Interventions: Drug: choline magnesium trisalicylate; Drug: Dexamethasone
- Choline Magnesium Trisalicylate (Experimental): Choline Magnesium Trisalicylate
  Interventions: Drug: choline magnesium trisalicylate

INTERVENTIONS:
Drug: choline magnesium trisalicylate — 1500mg orally every 8 hours beginning at hour 0 and continuing until hour 48.
Drug: Dexamethasone — 10mg orally every 6 hours beginning at hour 0 and continuing until hour 48.
  Arms: Dexamethasone plus Choline Magnesium Trisalicylate

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in cancer cells. It may also help doctors understand how cancer cells respond to treatment with choline magnesium trisalicylate.

PURPOSE: This pilot clinical trial is studying gene expression in cancer cells during chemotherapy and the safety of choline magnesium trisalicylate in treating patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine temporal changes in leukemic cell NF-kB activity when choline magnesium trisalicylate is administered during induction chemotherapy in patients with newly diagnosed acute myeloid leukemia.
* Determine toxicities of this regimen in these patients.

Secondary

* Determine patterns of leukemic cell gene expression in patients treated with this regimen.
* Determine if NF-kB modulation results in enhanced apoptosis in patients treated with this regimen.

OUTLINE: This is an open-label, pilot study.

Patients receive oral choline magnesium trisalicylate every 8 hours for 48 hours or dexamethasone every 6 hours for 48 hours plus choline magnesium trisalicylate every 8 hours for 48 hours during induction chemotherapy as determined by the primary physician.

Blood is collected at baseline, 24 hours, and 48 hours to assess for changes in NF-kB expression, apoptosis, and gene expression in leukemic cells.

PROJECTED ACCRUAL: A total of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed acute myeloid leukemia

  * Newly diagnosed disease
* Presence of cytogenetic abnormalities must be determined by standard cytogenetics with or without FISH studies
* Leukemic blast count > 5,000/mm³ of peripheral blood
* No acute promyelocytic leukemia (M3)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Bilirubin < 2.0 times upper limit of normal (ULN)
* AST < 3.0 times ULN
* Creatinine < 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled psychiatric illness that, in the opinion of the principal investigator, would preclude study compliance
* No other concurrent medical condition that would preclude study compliance
* No allergies to any investigational drugs and/or chemotherapeutic agents
* No upper or lower gastrointestinal (GI) related hemorrhage within the past 6 months as determined by endoscopy

  * No clinical diagnosis of GI bleeding requiring blood transfusions

PRIOR CONCURRENT THERAPY:

* No prior induction therapy
* No prior chemotherapy for acute leukemia
* No concurrent medications that would preclude study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Temporal changes in leukemic cell NF-kB activity | 5 years

SECONDARY OUTCOMES:
Patterns of leukemic cell gene expression after administration of choline magnesium trisalicylate | 5 years
Apoptosis related to NF-kB modulation | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

REFERENCES:
- [Result] Strair RK, Gharibo M, Schaar D, Rubin A, Harrison J, Aisner J, Lin HC, Lin Y, Goodell L, Anand M, Balsara B, Dudek L, Rabson A, Medina DJ. Nuclear factor-kappaB modulation in patients undergoing induction chemotherapy for acute myelogenous leukemia. Clin Cancer Res. 2008 Nov 15;14(22):7564-8. doi: 10.1158/1078-0432.CCR-08-1390. PMID 19010875